CLINICAL TRIAL: NCT01208051
Title: Phase I/II Trial of Cediranib Alone or Cediranib and Lenalidomide in Iodine 131-Refractory Differentiated Thyroid Cancer
Brief Title: Cediranib Maleate With or Without Lenalidomide for the Treatment of Thyroid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02530; NCI-2011-02530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-182-B; CDR0000685236; 10-182; P8317_A23PAMDREVW02; UCCRC-10-182-B; 8317 (Other: University of Chicago Comprehensive Cancer Center); 8317 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); N01CM00100 (NIH); N01CM62201 (NIH); P30CA014599 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Refractory Differentiated Thyroid Gland Carcinoma; Refractory Thyroid Gland Follicular Carcinoma; Refractory Thyroid Gland Hurthle Cell Carcinoma; Refractory Thyroid Gland Papillary Carcinoma; Unresectable Thyroid Gland Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid cancer, Hurthle cell; Thyroid Cancer, Papillary | interventions — cediranib; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Phase 1 was dose finding. Phase 2 parallel group comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (cediranib maleate) (Experimental): Patients receive cediranib maleate 30 mg PO QD on days 1-28. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis
- Arm B (cediranib maleate plus lenalidomide thru April 10, 2015) (Experimental): Patients receive cediranib maleate 30 mg PO and lenalidomide 15 mg PO on days 1-21. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. NOTE: As of April 10, 2015, patients assigned to this arm are discontinued lenalidomide and continued on cediranib alone.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Cediranib — Given PO
  Other Names: AZD2171
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm B (cediranib maleate plus lenalidomide thru April 10, 2015)

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of cediranib maleate when given together with or without lenalidomide and to see how well they work in treating patients with thyroid cancer. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stop the growth of thyroid cancer by blocking blood flow to the tumor. It is not yet known whether cediranib maleate is more effective when given together with lenalidomide in treating thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of cediranib maleate (cediranib) plus lenalidomide. (Phase I) II. Determine the progression-free survival rates of single agent cediranib in patients with iodine refractory, unresectable differentiated thyroid cancer (DTC) who have evidence of disease progression within 12 months of study enrollment. (Phase II) III. Determine the progression-free survival rates of cediranib in combination with lenalidomide in patients with iodine refractory, unresectable DTC who have evidence of disease progression within 12 months of study enrollment. (Phase II) IV. Compare the progression-free survival curves of single agent cediranib to combination therapy with cediranib with lenalidomide. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the response rate of cediranib in combination with lenalidomide in patients with iodine refractory, unresectable DTC who have evidence of disease progression within 12 months of study enrollment. (Phase I) II. Determine the toxicity, duration of response, progression free survival, and overall survival in patients with DTC treated with cediranib plus lenalidomide. (Phase I) III. Determine response rates and duration of response, early tumor size changes, the toxicity, and overall survival in patients with DTC treated with cediranib or cediranib plus lenalidomide. (Phase II) IV. Determine whether the presence of v-raf murine sarcoma viral oncogene homolog B1 (B-RAF) or V-Ki-ras2 Kirsten rat sarcoma (K-RAS) mutations in patients with DTC predict response to cediranib or cediranib plus lenalidomide. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Phase I: Patients receive cediranib maleate orally (PO) once daily (QD) on days 1-28 and lenalidomide PO QD on days 1-21 or 1-28. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Phase II: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive cediranib maleate PO QD on days 1-28. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive cediranib maleate PO and lenalidomide PO as in Phase I. NOTE: As of April 10, 2015, patients assigned to this arm are to discontinue lenalidomide and may continue on cediranib alone.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary, follicular, papillary/follicular variant or Hurthle cell carcinoma; patients must be felt to be poor candidates for or refractory to further surgery or radioactive I-131 therapy; I-131 therapy must have been completed at least 4 weeks prior to enrollment; all patients are expected to be on thyroxine suppression therapy
* Patients must have radiographically measurable disease; radiographically measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; lesions in previously irradiated anatomic areas (external beam radiation) cannot be considered target lesions unless there has been documented growth of those lesions after radiotherapy
* Patients must have evidence of disease progression (20% objective growth of existing tumors by Response Evaluation Criteria in Solid Tumors [RECIST] criteria) within the last 12 months
* In the Phase I portion, there is no limit on prior systemic therapies (cytotoxic or targeted therapies); however, patients who have discontinued previous vascular endothelial growth factor (VEGF) inhibitors secondary to adverse events are not eligible; in the Phase 2 portion, patients cannot have received more than 1 prior chemotherapy (cytotoxic or targeted) regimen; prior VEGF-pathway inhibitors or B-RAF inhibitors are permissible
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky > 60%)
* Leukocytes > 3,000/mcL
* Absolute neutrophil count (ANC) > 1,500/mcL
* Platelets > 100,000/mcL
* Hemoglobin > 9 g/dL
* Serum calcium < 12.0 mg/dL
* Total serum bilirubin below or equal to upper limit of institutional normal

  * Patients with hyperbilirubinemia due to Gilbert's syndrome may enroll in the trial
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine below or equal to upper limit of institutional limits OR creatinine clearance > 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have corrected QT interval (QTc) < 480 msec
* The following groups of patients are eligible provided that they have New York Heart Association (NYHA) class II cardiac function on baseline echocardiogram (ECHO)/multi-gated acquisition scan (MUGA):

  * Those with a history of class II heart failure who are asymptomatic on treatment
  * Those with prior anthracycline exposure
  * Those who have received central thoracic radiation that included the heart in the radiotherapy port
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Females of childbearing potential (FCBP) who receive cediranib alone must also have a negative initial and ongoing pregnancy tests as described above; FCBP who receive cediranib alone must also commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking cediranib; men on cediranib alone must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients receiving cediranib alone must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; at least 4 weeks must have elapsed since any major surgery; patients with prior use of thalidomide or lenalidomide are excluded
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; Note well (N.B): Patients with brain metastases with stable neurologic status following local therapy (surgery or radiation) for at least 8 weeks from definitive therapy and without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events are eligible for participation
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib, lenalidomide, or other agents used in this study
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) are ineligible
* Patients with 1+ or greater proteinuria on urinalysis should collect a 24 hour urine collection; patients with greater than 1.5 gram protein/24 hours are excluded
* Because lenalidomide may increase the risk of deep vein thrombosis (DVT) or pulmonary embolism (PE), patients must stop Epogen (epoetin alfa) at least 4 weeks prior to enrollment
* Patients with any condition (e.g., gastrointestinal tract disease resulting in malabsorption, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to absorb cediranib tablets or lenalidomide capsules are excluded; however, for patients who are unable to swallow cediranib tablets, cediranib tablets may be administered as a dispersion in water (ie, either drinking water, sterile water [for injection] or purified water); cediranib can be administered via nasogastric tube or gastrostomy tube; for patients unable to swallow lenalidomide whole, lenalidomide can be administered via gastrostomy feeding tube
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
  * Class III or IV heart failure as defined by the NYHA functional classification system
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illnesses/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study because cediranib and lenalidomide are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cediranib or lenalidomide, breastfeeding should be discontinued if the mother is treated with cediranib with or without lenalidomide
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cediranib or cediranib with lenalidomide; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yi Liao, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (33):
- United States (30):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center P2C, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology PA-Minneapolis, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 0: Cediranib 20 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (21/28 days, i.e., given for 15 days of a 28 day cycle)
- Phase I Dose Level +1: Cediranib 30 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (21/28 days, i.e., given for 21 days of a 28 day cycle)
- Phase I Dose Level +2: Cediranib 30 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (28/28 days, i.e., given for 28 days of a 28 day cycle)
- Phase II Arm A (Cediranib Maleate): Patients receive cediranib maleate 30 mg PO QD on days 1-28. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015): Patients receive cediranib maleate 30 mg PO and lenalidomide 15 mg PO on days 1-21. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. NOTE: As of April 10, 2015, patients assigned to this arm are discontinued lenalidomide and continued on cediranib alone.
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
Period: Total Enrollment
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
Started | 4 | 7 | 6 | 39 | 71
Completed | 4 | 6 | 5 | 39 | 69
Not Completed | 0 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 2
Not completed — Brain metastases | 0 | 0 | 1 | 0 | 0
Period: Interim Futility Analysis
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
Started | 0 | 0 | 0 | 39 | 68
Completed | 0 | 0 | 0 | 39 | 68
Not Completed | 0 | 0 | 0 | 0 | 0
Period: After Crossover to Cediranib Only
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
Started | 0 | 0 | 0 | 39 | 69 (One patient entered while futility analysis was ongoing.)
Completed | 0 | 0 | 0 | 39 | 69
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015) | Total
Number analyzed (Participants) | 4 | 6 | 5 | 39 | 69 | 123
Age, Continuous [Mean (Full Range); unit: years] | 72.2 [57 to 85] | 64.5 [55 to 78] | 67.2 [58 to 76] | 61.9 [27 to 86] | 63.8 [24 to 83] | 63.1 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 24 | 40 | 75
  Male | 0 | 2 | 2 | 15 | 29 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 3 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 5 | 2 | 7
  White | 4 | 6 | 4 | 30 | 59 | 103
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 5 | 7 | 12
  United States | 4 | 6 | 5 | 34 | 62 | 111

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Dose limiting toxicity was defined as any of the following occurring during the first cycle (28 days) of therapy:
  Hematological toxicities:
  * Any grade 4 neutropenia (ANC < 500) lasting more than 5 days
  * Any grade 4 neutropenia with concomitant fever (temperature > 38.5)
  * Any grade 4 neutropenia and sepsis or other severe infection
  * Any grade 4 thrombocytopenia
  Any other grade 3-4 non-hematological adverse drug reactions, except untreated nausea/vomiting, or hypersensitivity reactions.
  Grade 4 hypertension
  Grade 4 proteinuria Delay in the administration of a subsequent dose of cediranib and lenalidomide exceeding 2 weeks, due to an adverse drug reaction
Time Frame: 28 days
Population: Dose limiting toxicity was no an endpoint for the phase II study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
Number analyzed (Participants) | 4 | 6 | 5 | 0 | 0
Participants | 0 | 1 | 2 |  |

2. Primary Outcome: Progression-free Survival (Phase II Futility Analysis)
Description: Time from enrollment on study to disease progression or death from any cause. Surviving patients without progression are censored as of the date of the last negative examination. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. This analysis corresponds to the planned futility analysis after 40 events.
Time Frame: Assessed up to 3 years
Population: Phase I study did not have a futility analysis. For phase II, one patient in Arm B was enrolled while the futility analysis was ongoing.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 68
months |  |  |  | 20.9 [10.9 to NA] — Upper limit not reached, too few events | 10.6 [7.3 to 14.6]
Statistical Analysis 1: Comparison: Phase II Arm A (Cediranib Maleate) vs Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015); Test type: Superiority; p = 0.26, Log Rank — p-value is stratified by randomization factors; The conditional power was 7.8%, reaching the futility boundary of <15%. Patients on the combination arm were then crossed over to cediranib alone

3. Primary Outcome: Progression-free Survival (Final Results After Crossover)
Description: Time from study enrollment until disease progression or death from any cause. Surviving patients without progression are censored as of the date of the last negative examination. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Level 0: Cediranib 20 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (21/28 days, i.e., given for 15 days of a 28 day cycle)
- Dose Level +1: Cediranib 30 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (21/28 days, i.e., given for 21 days of a 28 day cycle)
- Dose Level +2: Cediranib 30 mg (28/28 days, i.e., given for 28 days of a 28 day cycle) + Lenalidomide 15 mg (28/28 days, i.e., given for 28 days of a 28 day cycle)
- Phase II Arm B (Cediranib Maleate Plus Lenalidomide): Patients receive cediranib maleate 30 mg PO and lenalidomide 15 mg PO on days 1-21. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. NOTE: As of April 10, 2015, patients assigned to this arm are discontinued lenalidomide and continued on cediranib alone.
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
Arm/Group | Dose Level 0 | Dose Level +1 | Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 4 | 6 | 5 | 39 | 69
months | NA [NA to NA] — Median not reached, too few events | 14.8 [3.5 to 30.9] | 23.6 [2.5 to 49.5] | 14.8 [8.5 to 23.8] | 11.3 [8.7 to 18.9]
Statistical Analysis 1: Comparison: Phase II Arm A (Cediranib Maleate) vs Phase II Arm B (Cediranib Maleate Plus Lenalidomide); Test type: Superiority; p = 0.36, Log Rank

4. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 | Dose Level +1 | Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 4 | 6 | 5 | 39 | 69
Participants | 0 | 2 | 4 | 17 | 30

5. Secondary Outcome: Overall Survival (Final Results After Crossover)
Description: Time from randomization to death from any cause. Patients who have not died are censored as of the date last known alive.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 0 | Dose Level +1 | Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 4 | 6 | 5 | 39 | 69
percentage of participants | NA [NA to NA] — 24 mo estimate not reached, too few events | 60.0 [17.1 to 100] | 100 [73.5 to 100] | 64.8 [43.3 to 86.4] | 75.3 [59.4 to 91.0]
Statistical Analysis 1: Comparison: Phase II Arm A (Cediranib Maleate) vs Phase II Arm B (Cediranib Maleate Plus Lenalidomide); Test type: Superiority; p = 0.80, Log Rank

6. Secondary Outcome: Percent Change in Tumor Size (Phase II)
Description: The percent change in tumor size from baseline to the end of cycle 2 (two months). The post-treatment total sum of lengths for a patient with a new lesion at cycle 2 will be scored as 1.2*max(pre-sum, post-sum) to ensure that the appearance of new lesions corresponds to a disease progression per Response Evaluation Criteria in Solid Tumors criteria. In the event of any early deaths prior to cycle 2, a nonparametric rank sum test will be used with deaths ranked at the extreme end of the distribution.
Time Frame: From baseline to 2 months
Population: Percent change in tumor size was not an endpoint for the phase I study.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Phase I Dose Level 0 | Dose Level +1 | Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 0 | 0 | 0 | 38 | 63
percent change |  |  |  | -12.5 [-26.0 to 0.0] | -4.2 [-25.0 to 0.0]
Statistical Analysis 1: Comparison: Phase II Arm A (Cediranib Maleate) vs Phase II Arm B (Cediranib Maleate Plus Lenalidomide); Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Serial Measurements of Thyroid Stimulating Hormone and Thyroglobulin
Description: Thyroid stimulating hormone and thyroglobulin levels
Time Frame: Up to 3 years
Population: These outcomes were not assessed in the Phase I study. These data were not collected and analyzed for the phase II study because combination treatment was stopped due to reaching futility criteria at interim analysis.
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Presence or Absence of B-RAF and RAS Mutations and Outcomes
Description: Presence or absence of B-RAF and RAS mutations at baseline--to be correlated with response rates, progression-free survival, and overall survival.
Time Frame: Up to 3 years
Population: Mutations were not endpoints for the phase I study. These data were not collected and analyzed in the phase II study because combination treatment was stopped due to reaching futility criteria at interim analysis.
Arm/Group | Dose Level 0 | Dose Level +1 | Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level +1 | Phase I Dose Level +2 | Phase II Arm A (Cediranib Maleate) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/5 | 8/39 | 13/69
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/6 | 5/5 | 16/39 | 32/69
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 5/5 | 38/39 | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0 (N=4) | Phase I Dose Level +1 (N=6) | Phase I Dose Level +2 (N=5) | Phase II Arm A (Cediranib Maleate) (N=39) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015) (N=69)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Blood bilirubin increase (Investigations) | 0 | 0 | 0 | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Death NOS (General disorders) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 5
Ejection fraction decreased (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Endocrine disorders - Other (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Neoplasms benihn, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Pain (General disorders) | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Social circumstances - Other (Social circumstances) | 0 | 0 | 0 | 1 | 0
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0 (N=4) | Phase I Dose Level +1 (N=6) | Phase I Dose Level +2 (N=5) | Phase II Arm A (Cediranib Maleate) (N=39) | Phase II Arm B (Cediranib Maleate Plus Lenalidomide Thru April 10, 2015) (N=69)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 6 | 10
Alanine aminotransferase increased (Investigations) | 2 | 5 | 3 | 12 | 31
Alkaline phosphatase increased (Investigations) | 2 | 2 | 1 | 6 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 10 | 18
Anorexia (Metabolism and nutrition disorders) | 4 | 4 | 5 | 22 | 31
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 6 | 8
Aspartate aminotransferase increased (Investigations) | 2 | 5 | 2 | 12 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 10 | 8
Blood bilirubin increased (Investigations) | 1 | 4 | 0 | 4 | 9
Blurred visioin (Eye disorders) | 0 | 0 | 0 | 1 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 12 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 8 | 16
Creatinine increase (Investigations) | 0 | 0 | 1 | 5 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 5 | 5 | 32 | 57
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 6 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 8 | 17
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 6 | 18
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 3 | 10
Eye disorders - Other (Eye disorders) | 0 | 0 | 0 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Fatigue (General disorders) | 4 | 6 | 5 | 31 | 57
Fever (General disorders) | 0 | 0 | 0 | 4 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 6
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 8
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 11 | 20
Hematuria (Renal and urinary disorders) | 0 | 3 | 2 | 5 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 8 | 11
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 5 | 4 | 6 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6 | 2
Hypertension (Vascular disorders) | 1 | 3 | 0 | 27 | 44
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 8 | 17
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 11 | 17
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 11 | 20
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 6
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 8 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2 | 9
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 2
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 2 | 6
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 6
Investigations - Other (Investigations) | 0 | 0 | 0 | 4 | 3
Lymphocyte count decreased (Investigations) | 2 | 0 | 3 | 7 | 12
Malaise (General disorders) | 0 | 0 | 0 | 2 | 2
Mood alteration-depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Mucositis oral (Gastrointestinal disorders) | 4 | 6 | 4 | 11 | 28
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 6 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 4
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 17 | 30
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 7
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 0 | 4 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 0 | 0 | 4 | 6
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 3 | 30
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 4 | 4
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 7
Pain (General disorders) | 1 | 1 | 1 | 11 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5 | 7
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 15 | 17
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 5 | 1
Platelet count decreased (Investigations) | 2 | 3 | 3 | 6 | 25
Proteinuria (Renal and urinary disorders) | 2 | 5 | 2 | 18 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 7
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 8 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 4 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 14 | 14
Weight loss (Investigations) | 0 | 0 | 1 | 16 | 20
White blood cell decreased (Investigations) | 2 | 2 | 3 | 3 | 28
Flu like symptoms (General disorders) | 0 | 0 | 0 | 2 | 1
CD4 lymphocytes decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 1 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 0
Salivary duct inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01208051/Prot_SAP_000.pdf